CLINICAL TRIAL: NCT05284084
Title: Prevention of Broncho-aspiration (BA) in Adult Subjects During Their ICU Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Juan Sanabria, Professor of Surgery, Vice-Chair & Scientific Director, Marshall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 945673-7
Record Dates: First submitted 2021-08-18; First posted 2022-03-17 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Bronchial Aspiration
Keywords: Bronchial; Aspiration; Bronchoaspiration; Broncho-aspiration; ICU; Intensive Care Unit; Surgical patients; Surgery
MeSH Terms: interventions — Histamine H2 Antagonists; Mouthwashes; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Negative Control (Placebo Comparator): Matched subjects by age, sex and BMI with no BA events, from a pool of 20,032 admission (01JAN2010 to 31DEC2019).
  Interventions: Other: Data collection for comparison
- Positive Control (Active Comparator): Matched subjects by age, sex and BMI with BA events, from a pool of 20,032 admission (01JAN2010 to 31DEC2019).
  Interventions: Other: Data collection for comparison
- Experimental group (Experimental): Consecutive subjects admitted to the ICU (these subjects will be matched with historical controls with and without BA events) from 30MAR2021 to 30MAR2022 on three subgroups:
  * Head up from the bed 15 degrees + H2 blockers + mouth wash BID
  * Head up from the bed 30 degrees + H2 blockers + mouth wash BID
  * Head up from the bed 45 degrees + H2 blockers + mouth wash BID
  Interventions: Other: Bed Head elevation, H2 blockers and mouth wash

INTERVENTIONS:
Other: Bed Head elevation, H2 blockers and mouth wash — Elevation of the bed head to 15, 30 and 45 degrees, daily H2 blockers administration and mouth wash BID.
  Arms: Experimental group
Other: Data collection for comparison — Data collection for comparison
  Arms: Negative Control; Positive Control

SUMMARY:
Patients of age >18 yo, admitted to the ICU through the surgery department from 2AUG2021 to 1AUG2022 will be divided into three groups:

1. Patients admitted to the ICU in the first 3-4 months will have their bed head elevated to 15 degrees + H2 blockers administration + mouth wash BID
2. Patients admitted to the ICU in the following 3-4 months will have their bed head elevated to 30 degrees + H2 blockers administration + mouth wash BID
3. Patients admitted in the last 3-4 months will have their bed head elevated to 45 degrees + H2 blockers administration + mouth wash BID.

All patients will have their vital signs, BMI, and fluids ins and outs measured every 24 hours until the discharge from the ICU or death. All patients will be evaluated for GI functions (no vomiting, flatus+, bowel movement +, bowel sounds+, and KUB with normal gas distribution pattern) prior to oral intake.

Patients in the three groups will be matched by age, sex, and BMI with historical controls with broncho- aspiration (BA) (positive controls) and without BA events (negative controls) from a pool of 20,032 ICU admissions (01JAN2010 to 31DEC2019).

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* All the patients admitted to ICU by surgery department.
* Development of aspiration pneumonia in patients admitted to ICU department of VA hospital.
* Aspiration Pneumonia development during hospital stay and treating physician indicated the diagnosis of aspiration pneumonia in history and physical exam notes.

Exclusion Criteria:

* Age <18
* Patient transferred or admitted to the hospital as a primary diagnosis of aspiration pneumonia (development of aspiration pneumonia prior to admission).
* Treating physician not documented aspiration pneumonia in history or physical exam notes.
* Drug overdose, seizure or cardiopulmonary arrest prior to hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Rate of Bronchospiration pneumonia among study participants during their ICU admission | 12 Months
  Calculating the number of subjects who developed bronchoaspiration pneumonia compared to the total number of ICU admission

SECONDARY OUTCOMES:
Determine if there is an association between BA events and death rate in the ICU for the specified time period | 12 Months
  Determining the factors impacting the rate of bronchaspiration and the rate of related death

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanabria, MD MSc FACS, Principal Investigator — Marshall University School of Medicine
Locations (1):
- Marshall University School of Medicine, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No